CLINICAL TRIAL: NCT05373680
Title: Clinical Study Evaluating the Efficacy and Safety of Metformin Versus Empagliflozin for Halting Chronic Kidney Disease Progression
Brief Title: Efficacy and Safety of Metformin Versus Empagliflozin on Chronic Kidney Disease Progression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Bassant Maher Mahboub, Principal Investigator: Bassant Maher Abbas Mahboub, PhD candidate., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34976/10/21
Record Dates: First submitted 2022-02-18; First posted 2022-05-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2023-04

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Metformin; Empagliflozin; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Metformin; Biguanides; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Metformin treatment group (Experimental): In this arm, patients with chronic kidney disease who meet study inclusion criteria will receive metformin 1000 mg PO daily added to their usual therapy.
  Interventions: Drug: Metformin; Other: Control
- Empagliflozin treatment group (Experimental): In this arm, patients with chronic kidney disease who meet study inclusion criteria will receive empagliflozin 10 mg daily PO added to their usual therapy.
  Interventions: Drug: Empagliflozin; Other: Control
- Control group (Other): In this arm, patients with chronic kidney disease who meet study inclusion criteria will receive their usual therapy.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Metformin — Patients will receive metformin 1000 mg PO daily added to their usual therapy for the management of CKD (including the management of predisposing causes with other supportive care).
  Other Names: Biguanide
  Arms: Metformin treatment group
Drug: Empagliflozin — Patients will receive empagliflozin 10 mg daily PO added to their usual therapy for the management of CKD (including the management of predisposing causes with other supportive care).
  Other Names: Sodium glucose cotransporter-2 (SGLT2) inhibitor
  Arms: Empagliflozin treatment group
Other: Control — Patients will receive their usual therapy for the management of CKD (including the management of predisposing causes with other supportive care).

SUMMARY:
This randomized controlled trial aims at evaluating the efficacy and safety of the antidiabetics metformin versus empagliflozin on chronic kidney disease (CKD) progression in patients with CKD stages 2 or/and 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild or/and moderate chronic kidney disease (stages 2 or/and 3, estimated glomerular filtration rate (eGFR) between 30-89 ml/min/1.73 m2) at the time of the baseline visit.
* Patients with and without type 2 diabetes.
* Patients with or without proteinuria.
* Age: ≥ 18 years.

Exclusion Criteria:

* Type 1 diabetes.
* Patients with eGFR ˂30 ml/min/1.73 m2.
* Patients with known hepatic cell failure.
* Decompensated heart requiring acute management.
* Active malignancy.
* Planned coronary or surgical interventions.
* Known hypersensitivity to study medications.
* Chronic inflammation, trauma, or infection.
* Pregnant or lactating women.
* Patients already on metformin or a sodium-glucose cotransporter-2 (SGLT2) inhibitor.
* Any of the study treatments labeled contraindications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) values from baseline | Period of 12 months
  This will be achieved by measuring the serum creatinine levels and then eGFR values will be calculated.

SECONDARY OUTCOMES:
Change in albumin or protein excretion values from baseline | Period of 12 months
  This will be achieved by measuring the urinary albumin or protein:creatinine ratio from a spot urine test in a morning sample.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mansoura University, Al Mansurah, Dakahlia Governorate
  - Tanta University Teaching Hospitals, Tanta, Gharbia Governorate

REFERENCES:
- [Derived] Mahboub BM, Refaie AF, El-Haggar SM, Hafez YM, Mostafa TM. Efficacy and safety of metformin versus empagliflozin on chronic kidney disease progression (MET-EMPA-CKD): a randomized controlled trial. Diabetol Metab Syndr. 2025 Dec 10;18(1):17. doi: 10.1186/s13098-025-02040-9. PMID 41373013
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240